CLINICAL TRIAL: NCT04708691
Title: Effects of Aerobic Exercise Modulation on Brain Physiology and Cognition
Brief Title: Effects of Aerobic Exercise Modulation on Brain Physiology and Cognition in Young Adults With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201911100RIND
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-05

CONDITIONS: Depression
Keywords: Depression; Neurophysiology; Cognition
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): aerobic exercise for 30 mins
  Interventions: Other: Aerobic exercise
- Control (No Intervention): sitting for 30 mins

INTERVENTIONS:
Other: Aerobic exercise — aerobic exercise
  Arms: Aerobic exercise

SUMMARY:
Major depressive depression (MDD) affects a quarter of young adults and is associated with marked global burden in this population. Recently, growing literature has shown that cognitive dysfunction is common in young adults with depression. There is a vast amount of evidence indicating aerobic exercise has positive effects on cognitive function in healthy as well as in subjects with depression. The results might be dependent on neuroplastic changes induced by aerobic exercise. Nevertheless, the neurocognitive mechanisms of aerobic exercise in young adults with depression has not received systematic investigation. In addition, the association between the underlying brain physiology and cognitive performance has not been explored so far. In this project, the investigators aim to explore the relevance of a single session of aerobic exercise for human brain physiology and the impact of respective physiological effects on cognitive processes in young adults with depression.

DETAILED DESCRIPTION:
The study are interested in the physiological foundation of the impact of aerobic exercise on cognitive performance in youth MDD subjects. Combined application of neurophysiological intervention and recording tools, including non-invasive brain stimulation, is suited to explore the impact of aerobic exercise on brain physiology and cognition in humans. We will apply transcranial magnetic stimulation (TMS) to obtain evoked potentials with electromyography (EMG) to explore cortical excitability. In the same participants, we will combine motor learning, working memory, and attention task to explore the association between the physiological effect of aerobic exercise and respective cognitive alterations. This project aims to explore the impact of aerobic exercise on cortical excitability and cognitive performance, and the association between these phenomena in youth MDD subjects. The study will improve our understanding of the role of aerobic exercise in cortical excitability, an important physiological basis for cognitive processes in humans, the underlying physiological mechanisms with regard to the aerobic exercise, and their functional relevance in youth MDD subjects.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of major depressive disorder by a board-certified psychiatrist according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
2. Total score of the 17-item Hamilton Rating Scale for Depression (HAM-D) less than 7
3. Aged between 18 to 35 years
4. Right handedness

Exclusion criteria

1. A major depressive episode within the past three months
2. Pacemaker or deep brain stimulation
3. Metal implants in the head or neck area
4. Other major mental disorders including autism spectrum disorders, mental retardation, psychotic disorders, bipolar disorders, obsessive-compulsive disorder, and neurocognitive disorders
5. Alcohol or other illicit substance abuse
6. Neurological diseases involving the central nervous system
7. Major debilitating systemic diseases
8. Pregnancy
9. Breast feeding
10. Cigarette smoker
11. Color blindness
12. Take part in another study within the last 4 weeks

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability | 4 weeks
  TMS measurment

SECONDARY OUTCOMES:
Cognitive task | 4 weeks
  Serial reaction time task, 3-back letter task

CONTACTS AND LOCATIONS:
Overall Officials: Kuo Hsiao-I, PHD, Principal Investigator — Assistant Professor, National Taiwan University; Kuo Hsiao-I, Principal Investigator — Assistant Professor, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan